CLINICAL TRIAL: NCT04792814
Title: Intraoperative Cell Salvage and Retrograde Autologous Priming in Patients Undergoing Isolated Coronary Bypass Grafting and Conventional Aortic Valve Replacement.
Brief Title: Cell Salvage and Retrograde Autologous Priming
Status: Completed | Type: Observational
Sponsor: University Hospital Schleswig-Holstein (Other)
Responsible Party: Principal Investigator, Dr. Jochen Renner, Prof. Dr. med. Jochen Renner, University Hospital Schleswig-Holstein
Other Study IDs: IN-MAT_RAP_01
Record Dates: First submitted 2020-12-17; First posted 2021-03-11 (Actual); Last update posted 2021-03-11 (Actual); Status verified 2021-03

CONDITIONS: Surgery; Hemodynamic Instability
Keywords: cell salvage; length of stay in hospital; mortality

STUDY DESIGN:
Observational Model: Case-Control | Time Perspective: Retrospective
Oversight: Data Monitoring Committee: No | FDA-regulated Drug: No | FDA-regulated Device: No

GROUPS / COHORTS (2):
- MAT-RAP group: MAT and RAP
- historical group: standard procedure

SUMMARY:
In recent years Patient Blood Management (PBM) has developed into a multifactorial and interdisciplinary concept that focuses on individualized and optimized hemotherapy. Of course, this also applies to the cardiac surgery area (1). In this context, the quality of the intraoperative PBM can be represented by patients scheduled for isolated coronary artery bypass grafting (CABG) and isolated aortic valve replacement (AVR). In a prospective, observational "before-and-after" protocol, the investigators analysed the impact of the combined use of retrograde autologous priming (RAP) and cell salvage on intraoperative usage of red blood cell concentrates (RBC) (2).

DETAILED DESCRIPTION:
200 patients (CABG or AVR) will be monitored using local standard of care in these patients without cell salvage and RAP (control group, CG), followed by 200 patients with cell salvage and RAP (study group, SG). Both groups are defined by elective surgery and hemodynamically stable patients prior to the onset of the cardiopulmonary bypass (CPB). Based on our own data and current data from the literature, the investigators assume that the use of MAT in combination with RAP leads to at least an intraoperative reduction of the erythrocyte consumption of 15%. Consequently, the investigators calculated a case number of approximately 200 patients per group.

The study is set up with a control group under previous standard therapy. The data is recorded and analyzed descriptively. Qualitative comparisons will be made in the discussion of previously published data.

ELIGIBILITY:
Inclusion Criteria:

* scheduled for cardiac surgery
* informed written consent

Exclusion Criteria:

* rejection by the patient
* switching to another procedure

Min Age: 18 Years | Sex: All | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Study Population: heart surgery patients (CABG and aortic valve replacement)
Sampling Method: Non-Probability Sample
Enrollment: 200 (Actual)
Dates: Start 2018-06-01 (Actual); Primary Completion 2019-10-31 (Actual); Study Completion 2019-10-31 (Actual)

PRIMARY OUTCOMES:
number of red blood cell concentrates | through study completion, an average of 1 year
  use of RBC

SECONDARY OUTCOMES:
postoperative complications | through study completion, an average of 1 year
  acute renal failure, pulmonary edema, pneumonia, wound infection
length of stay in hospital | through study completion, an average of 1 year
  time in hospital after surgery
hospital mortality | through study completion, an average of 1 year
  hospital mortality

CONTACTS AND LOCATIONS:
Overall Officials: Jochen Renner, Prof. Dr., Study Chair — UKSH, Campus Kiel
Locations (2):
- Germany (2):
  - Universitätsklinikum Schleswig-Holstein Campus Kiel - Klinik für Anästhesiologie und Operative Intensivmedizin, Kiel, Deutschland (deu)
  - GERMANY - Universitätsklinikum Schleswig-Holstein, Kiel, Schleswig-Holstein

IPD SHARING:
Plan to Share IPD: No

REFERENCES:
- [Background] Pagano D, Milojevic M, Meesters MI, Benedetto U, Bolliger D, von Heymann C, Jeppsson A, Koster A, Osnabrugge RL, Ranucci M, Ravn HB, Vonk ABA, Wahba A, Boer C. 2017 EACTS/EACTA Guidelines on patient blood management for adult cardiac surgery. Eur J Cardiothorac Surg. 2018 Jan 1;53(1):79-111. doi: 10.1093/ejcts/ezx325. No abstract available. PMID 29029100
- [Background] Meybohm P, Choorapoikayil S, Wessels A, Herrmann E, Zacharowski K, Spahn DR. Washed cell salvage in surgical patients: A review and meta-analysis of prospective randomized trials under PRISMA. Medicine (Baltimore). 2016 Aug;95(31):e4490. doi: 10.1097/MD.0000000000004490. PMID 27495095